CLINICAL TRIAL: NCT07123402
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-finding Phase II Clinical Trial to Evaluate the Efficacy and Safety of TRD205 Tablets in the Treatment of Chronic Postoperative Neuralgia
Brief Title: To Evaluate the Efficacy and Safety of TRD205 Tablets in the Treatment of Chronic Postoperative Neuralgia
Acronym: TRD205
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tide Pharmaceutical Co., Ltd (Industry)
Collaborators: China-Japan Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRD205-II-01
Record Dates: First submitted 2025-07-31; First posted 2025-08-14 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Chronic Postoperative Neuralgia
Keywords: chronic postoperative neuralgia; TRD205

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 200mg treatment group (Experimental): Take TRD205 tables or placebo orally once a day every morning for 6 consecutive weeks
  Interventions: Drug: TRD205 tablets
- 400mg treatment group (Experimental): Take TRD205 tables or placebo orally once a day every morning for 6 consecutive weeks
  Interventions: Drug: TRD205 tablets
- 600mg treatment group (Experimental): Take TRD205 tables or placebo orally once a day every morning for 6 consecutive weeks
  Interventions: Drug: TRD205 tablets
- Placebo (Placebo Comparator): Take placebo orally once a day every morning for 6 consecutive weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRD205 tablets — orally ;Take TRD205 1 tablets and Placebo 2 tablets
  Arms: 200mg treatment group
Drug: TRD205 tablets — orally ;Take TRD205 2 tablets and Placebo 1 tablets
  Arms: 400mg treatment group
Drug: TRD205 tablets — orally ;Take TRD205 3 tablets and Placebo 0 tablets
  Arms: 600mg treatment group
Drug: Placebo — orally ;Take Placebo 3 tablets
  Arms: Placebo

SUMMARY:
This is a phase II, multicenter ,randomized, double-blind, placebo-controlled, dose-finding study designed to evaluate the efficacy and safety of TRD205 tablets in the treatment of chronic postoperative neuralgia

DETAILED DESCRIPTION:
This study used a placebo as a control to explore the efficacy, safety and pharmacokinetic characteristics of multiple administration of TRD205 tablets at different doses forchronic postoperative neuralgia .

ELIGIBILITY:
Inclusion Criteria:

* 18 Years ≤ Age ≤ 80 years (calculated as time of signing ICF), both male and female.
* Subject experienced pain following surgical procedures including Thyroid gland and Breast surgery, orthopedic surgery , thoracotomy Etc. (except neurosurgery, amputation, cesarean section).
* Chronic pain ≥ 3 months post-op with pain localized to the operative site, Or The area of innervation that projects to the nerve at this site (Including radicular pain radiating to one side or limb after spinal surgery) Or involving the dermatome.
* DN4 scale ≥ 4, AND The subject's pain was judged by the investigator to be neuropathic in nature.
* Subjects had moderate to severe pain intensity (ie, averaged over the single-blind run-in period NRS Score ≥ 4 Points, see requirements for single-blind run-in period and randomization criteria for details).
* The subject is able to communicate well with the investigators, fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign the informed consent form .
* Subject is willing to voluntarily use the contraception specified in the protocol from signing the ICF to 1 month after the last dose of investigational drug (For details see Fig. 附录4) . Both male and female subjects had no plans to donate sperm or ova during the study and for 1 month after investigational product administration.

Exclusion Criteria:

* Investigator Judge the pain of subjects in whole or in part Pathological pain or pain in the central nervous system Caused by other postoperative complications (e.g., infection, disease recurrence, etc.).
* Present Other Causally induced pain, such as the presence of skin disease in the affected skin area, cervical and lumbar spine disease, trauma, etc., thus affecting the investigator's evaluation of CPSNP or confusing the subject's self-assessment of CPSNP.
* Presence of other neurological or psychiatric disorders that, in the judgment of the investigator, could confound the subject's self-assessment of CPSNP or affect the subject's ability to complete diary card completion.
* Known history of hypersensitivity to investigational products or components or excipients of rescue medication during the study period, or history of hypersensitivity to two or more drugs.
* Previously Received Any prohibited medication or non-drug therapy, and in Fig. Single-Blind Run-in Period Pre Did not undergo the protocol-required washout period (excluded medications Elution Phase: Single-Blind Run-in Period ≥ 5 half-lives or 7 days prior, whichever is longer; non-drug therapy is prohibited Elution Phase: Single-Blind Run-in Period ≥ 30 days prior) that may interfere with the evaluation of the test drug during the study.
* Have an electrical stimulation instrument or intrathecal drug infusion system implanted to treat pain.
* History of alcoholism (> 14 units/week of alcohol, 1 unit is equivalent to 360 mL of beer, or 45 mL of spirits with 40% alcohol, or 150 mL of wine) or drug abuse or drug abuse within 1 year prior to signing the ICF.
* Patients with clinically significant acute or chronic diseases or unstable diseases, such as but not limited to acute cardiovascular disease, cerebrovascular disease, liver, kidney, respiratory system, blood system, immune system and other diseases, inflammatory or rheumatic diseases, uncontrolled infection, untreated endocrine diseases, etc., and affecting the subjects at the investigator's discretion.
* Present Dysphagia Or any gastrointestinal disorder affecting drug absorption.
* Malignancy diagnosed within 2 years prior to signing the ICF (with the exception of non-metastatic cutaneous basal cell or squamous cell carcinoma or carcinoma in situ of the cervix that has been appropriately treated or excised).
* Patients with previous suicidal behavior or a positive response to Item 4 or 5 on the C-SSRS scale (for the 12 months prior to signing the ICF) .
* Systolic BP ≥ 160 mmHg and/or diastolic BP ≥ 100 mmHg; Systolic pressure ≤ 90 mmHg and/or diastolic pressure ≤ 60 mmHg; Heart rate < 50 or > 110 beats per minute.
* Neutrophil count < 1.5 × 10 9 /L; platelet count < 100 × 10 9 /L; Aspartate aminotransferase (AST) > 2.0 × upper limit of normal (ULN); alanine aminotransferase (ALT) > 2.0 × ULN; Urea or urea nitrogen (Urea or BUN) > 1.5 × ULN; Creatine kinase > 2.0 × ULN; Estimated serum creatinine clearance < 60 mL/min by Cockcroft-Gault formula.
* Treponema pallidum antibody or human immunodeficiency virus antibody positive in any test at screening and judged by the investigator as not suitable for the subject .
* Subjects who are expected to require reoperation from signing the ICF to the end of the study.
* Females who are lactating or pregnant, or intend to become pregnant (female subjects or partners of male subjects) during the study period and within 1 month after dosing.
* Those who have participated in or are participating in other clinical trials within 1 month prior to signing the ICF.
* Other conditions not suitable for inclusion as judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-05-27 (Estimated)

PRIMARY OUTCOMES:
The change in the weekly average NRS (numeric pain rating scale,0~10:0 equated to no pain, and 10 equated to the worst pain imaginable )pain score from baseline after 6 weeks of treatment | 8 weeks
  The Digital Assessment Scale (NRS) is used to evaluate the degree of pain in patients using the 11-point numeric pain rating scale (0-10; 0 equated to no pain, and 10 equated to the worst pain imaginable).The NRS pain score will be was assessed during the single-blind introduction period, the double-blind treatment period, and at the early end of the visit.The baseline of the NRS pain score is defined as the weekly average of the NRS pain score collected during the single-blind introduction period. Before taking the medicine every morning, the subjects retrospectively evaluated the average pain level in the past 24 hours. In addition, 1 hour before each remedial analgesia, the average pain intensity from the previous use of the investigational drug to the use of the remedial medication should be retrospectively assessed.NRS scores were collected at Visit 3, Visit 4, Visit 5, Visit 6, Visit 7, and at the early end of the visit for the calculation of the weekly average score.

SECONDARY OUTCOMES:
Treatment-Related Adverse Events | 7 weeks
  Assessment of all AEs, SAEs and TEAEs
Peak Plasma Concentration（Cmax） | Within 4 hours after the last administration
  Two samples were collected before administration at Visvisit 7( the last administration) and within 1 to 4 hours after administration.The blood drug concentration data of TRD205 obtained in this study will be combined with the previously completed clinical research data for population pharmacokinetic analysis (using the nonlinear mixed-effects model [NONMEM]), and a population pharmacokinetic model will be established to characterize the PK characteristics of TRD205.Then, based on the parameter estimates of the established final population pharmacokinetic model, the individual exposure parameters of the subjects were estimated for further dose-effect (exposing-effect) analysis, including the correlation exploration analysis of PK/ efficacy and PK/ safety.
Area under the plasma concentration versus time curve （AUC） | Within 4 hours after the last administration
  Two samples were collected before administration at Visvisit 7( the last administration) and within 1 to 4 hours after administration.The blood drug concentration data of TRD205 obtained in this study will be combined with the previously completed clinical research data for population pharmacokinetic analysis (using the nonlinear mixed-effects model [NONMEM]), and a population pharmacokinetic model will be established to characterize the PK characteristics of TRD205.Then, based on the parameter estimates of the established final population pharmacokinetic model, the individual exposure parameters of the subjects were estimated for further dose-effect (exposing-effect) analysis, including the correlation exploration analysis of PK/ efficacy and PK/ safety.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided